CLINICAL TRIAL: NCT06090864
Title: The Administration of T Lymphocytes Expressing the CD30 Chimeric Antigen Receptor (CAR) and CCR4 for Relapsed/Refractory CD30+ Hodgkin s Lymphoma
Brief Title: ATLCAR.CD30.CCR4 for CD30+ HL ATLCAR.CD30.CCR4 Cells
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2222-ATL
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin Lymphoma; Relapse; Refractory
Keywords: cellular therapy; CD30+
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Drug Therapy; Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATLCAR.CD30 (Experimental): Subjects will be enrolled on 1 of 3 dose levels as determined by a 3+3 design. Up to 25 evaluable subjects may then be enrolled in the phase II portion of the study. Subjects may have cells procured to manufacture the ATLCAR.CD30.CCR4 cells if they meet eligibility for procurement. During the time period necessary to manufacture the ATLCAR.CD30.CCR4 cells, Subjects will be allowed to receive standard-of-care bridging therapy at the discretion of their local oncologist. Prior to cell infusion, subjects will undergo additional eligibility evaluations, and then if eligible, will undergo lymphodepletion followed by cell infusion 2-14 days later. Subjects will then be followed for 15 years as is required for studies involving gene transfer experiments
  Interventions: Drug: Chemotherapy; Biological: Cell infusion

INTERVENTIONS:
Drug: Chemotherapy — Subjects will receive a lymphodepletion regimen of bendamustine 70 mg/m2 IV and fludarabine 30 mg/m2 each as a daily infusion for 3 consecutive days prior to the ATLCAR.CD30.CCR4 cell infusion.
Biological: Cell infusion — ATLCAR.CD30.CCR4 cells infusion for the eligible subjects after depletion chemotherapy.

SUMMARY:
Despite the progress in the therapy, Hodgkin's Lymphoma (HL) remains fatal for more than 15% of patients. Even in patients who are cured, the morbidity of therapy is substantial and long-lasting. New therapeutic agents are required therefore not only to further reduce mortality but also to alleviate morbidity.

The majority of HL express the CD30 antigens. CD30 expression is routinely used for the diagnosis of HL. Preclinical observations support CD30 as a viable target of CAR-T therapy. This phase Ib/II study was conducted based on these observations.

The purpose of this study is to determine the tolerability of ATLCAR.CD30.CCR4 cells in subjects with Hodgkin's Lymphoma and identify a recommended dose for further.

This is a single-center, open-label phase Ib/II trial that uses a 3+3 design to identify a recommended phase 2 dose (RP2D) of ATLCAR.CD30.CCR4 cells in Hodgkin's Lymphoma. The phase II portion is designed to determine the PFS of ATLCAR.CD30.CCR4 in Hodgkin's Lymphoma.

Subjects will be enrolled on 1 of 3 dose levels as determined by a 3+3 design. Up to 25 evaluable subjects may then be enrolled in the phase II portion of the study. Subjects may have cells procured to manufacture the ATLCAR.CD30.CCR4 cells if they meet eligibility for procurement. During the time period necessary to manufacture the ATLCAR.CD30.CCR4 cells, Subjects will be allowed to receive standard-of-care bridging therapy at the discretion of their local oncologist. Prior to cell infusion, subjects will undergo additional eligibility evaluations, and then if eligible, will undergo lymphodepletion followed by cell infusion 2-14 days later. Subjects will then be followed for 15 years as is required for studies involving gene transfer experiments.

ELIGIBILITY:
During the period of cell procurement and lymphodepletion, subjects will be eligible to receive standard-of-care therapy e.g., chemotherapy or radiation therapy to stabilize their disease if the treating physician feels it is in the subject's best interests. Eligibility must be maintained up until the subject is procured, receives lymphodepletion, or receives treatment for the subject to be considered eligible to proceed with the specific phase of the study.

Inclusion Criteria:

Unless otherwise noted, subjects must meet all of the following criteria to participate in all phases of the study. As these criteria are unchanging they will be evaluated at the time of initial enrollment and not continuously throughout the study.

1. Written informed consent and HIPAA authorization for release of personal health information explained to, understood by, and signed by the subject or legally authorized representative.
2. Age ≥ 18 years at the time of consent.
3. Karnofsky score of > 60%
4. The subject must have a diagnosis of Classical Hodgkin Lymphoma according to World Health Organization criteria.

Exclusion Criteria:

1. Subjects had major surgery within 28 days.
2. Subject received investigational agents or tumor vaccines within 3 weeks.
3. Subject received chemotherapy or radiation therapy within the previous 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b adverse events | Up to 6 weeks
  Toxicity will be graded as the number of participants with adverse events (AE) related to the administration of ATLCAR.CD30.CCR4 cells in subjects with CD30+ Hodgkin's Lymphoma.
  AEs will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Dose Limiting Toxicities (DLTs) are defined as at least possibly related to CAR.B7-H3T cell product administration.
Phase 1b Toxicity Cytokine Release Syndrome (CRS) | Up to 6 weeks
  CRS will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading related to the administration of ATLCAR.CD30.CCR4 cells in subjects with CD30+ Hodgkin's Lymphoma. Grade 1 - Mild: Fever ≥38^ o C, No hypotension, No hypoxia, Grade 2 - Moderate: Fever ≥38^ o C, Hypotension not requiring vasopressors, Hypoxia requiring low-flow nasal cannula (≤6 L/minute) or blow-by, Grade 3 - Severe: Fever ≥ 38^ o C, Hypotension requiring a vasopressor with or without vasopressin, Hypoxia requiring high-flow nasal cannula (>6 L/minute), facemask, nonrebreather mask, or Venturi mask, Grade 4 - Life-threatening: Fever ≥38^oC, Hypotension requiring multiple vasopressors (excluding vasopressin), Hypoxia requiring positive pressure (e.g. Continuous positive airway pressure, BiPAP, intubation, mechanical ventilation), Grade 5 - Death
Phase 1b Toxicity Immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 6 weeks
  Neurotoxicity will be graded according to the Immune effector cell-associated neurotoxicity syndrome (ICANS) criteria related to the administration of ATLCAR.CD30.CCR4 cells in subjects with CD30+ Hodgkin's Lymphoma.
  Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).
Phase II Median Progression Free Survival (PFS) | Up to 6 months
  Median PFS will be measured from the first day of lymphodepletion chemotherapy prior to ATLCAR.CD30.CCR4 cell infusion to progression (as defined by Lugano Criteria or death. Complete: Complete metabolic response on Positron emission tomography (PET) or the largest transverse diameter (LDi) of target nodes/masses ≤ 1.5 cm and no extra lymphatic disease on Computerized Tomography (CT). Partial: reduced uptake compared with baseline and residual mass(es) on PET and ≥50% decrease in the sum of the products of diameters (SPD) of nodes and extranodal sites on CT. No Response or Stable Disease: No metabolic response on PET or < 50% decrease from baseline in SPD, measurable nodes and extranodal sites; no criteria for the progressive disease are met on CT. Progressive Disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new focus on PET, LDi>1.5 cm or by ≥ 50% from nadir.

SECONDARY OUTCOMES:
Phase Ib Dose Limiting Toxicity | Up to 6 weeks
  The recommended phase 2 dose (RP2D) of ATLCAR.CD30.CCR4 cells will be determined based on the 3+3 dose finding rule as specified in the protocol for the tolerability of ATLCAR.CD30.CCR4 cells will be assessed using NCI-CTCAE v5 and ASTCT Consensus CRS Grading Criteria.
  * Grade 3-5 allergic reactions related to the CAR-T cell infusion.
  * A treatment-emergent Grade 3 CRS that does not improve to Grade 0-1 by 72 hours or Grade 4 CRS
  * Grade ≥3 ICANS that are unresponsive to the standard of care interventions and do not decrease to Grade ≤1 within 7 days or grade 4 ICANS of any duration that has evidence of cerebral edema and/or generalized convulsive status epilepticus.
  * Any treatment-emergent Grade 4 non-hematologic AE that does not resolve to Grade 2 within 7 days.
  * Any Grade 5 events are not due to the underlying malignancy.
Overall Survival (OS) | Up to 6 months
  OS is defined as the time from the first day of lymphodepletion to date of death for any cause. Subjects who have not had an event will be censored at the date of last assessment documenting the subject was alive.
Duration of Response (DOR) | Up to 6 months
  DOR is defined as the time from partial response (PR) or better to progressive disease (PD) per Lugano Criteria. Complete Response: Complete metabolic response on Positron emission tomography (PET) or Target nodes/nodal masses must be ≤ 1.5 cm in the largest transverse diameter (LDi) or no extra lymphatic of disease on Computerized Tomography (CT). Partial Response: Score of 4 or 5† with reduced uptake of any size on PET and ≥50% decrease in the sum of the products of diameters (SPD) of nodes and extranodal sites on CT. No Response or Stable Disease: No metabolic response on PET or < 50% decrease from baseline in SPD of nodes and extranodal sites; no criteria for the progressive disease are met on CT. Progressive Disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials